CLINICAL TRIAL: NCT06524674
Title: A Single-Blind, Controlled, Cross-Over Clinical Study to Compare the Effect of an Oral Rehydration Solution on the Rate of Absorption of Functional Ingredients
Brief Title: Clinical Study to Compare the Effect of an Oral Rehydration Solution on the Rate of Absorption of Functional Ingredients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liquid I.V. (Other)
Collaborators: Princeton Consumer Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PKPD
Record Dates: First submitted 2024-06-11; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Absorption; Pharmacokinetic
MeSH Terms: interventions — Sleep

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sleep (Active Comparator): Participants self-administered one serving of an oral rehydration solution followed by subsequent blood draws
  Interventions: Dietary Supplement: Hydration Multiplier + Sleep
- Energy (Active Comparator): Participants self-administered one serving of an oral rehydration solution followed by subsequent blood draws
  Interventions: Dietary Supplement: Hydration Multiplier + Energy
- Sleep Comp (Placebo Comparator): Participants self-administered one serving of an oral rehydration solution followed by subsequent blood draws
  Interventions: Other: Sleep Comp
- Energy Comp (Placebo Comparator): Participants self-administered one serving of an oral rehydration solution followed by subsequent blood draws
  Interventions: Dietary Supplement: Energy Comp

INTERVENTIONS:
Dietary Supplement: Hydration Multiplier + Energy — Participants will be administered one oral serving of an oral rehydration solution containing caffeine and l-theanine
  Arms: Energy
Dietary Supplement: Hydration Multiplier + Sleep — Participants will be administered one oral serving of an oral rehydration solution containing melatonin and l-theanine
  Arms: Sleep
Dietary Supplement: Energy Comp — Participants will be administered one oral serving of a comparator oral rehydration solution containing caffeine and l-theanine
  Arms: Energy Comp
Other: Sleep Comp — Participants will be administered one oral serving of a comparator oral rehydration solution containing melatonin and l-theanine
  Arms: Sleep Comp

SUMMARY:
The objective of this study was to compare the individual pharmacokinetics of functional ingredients included in an oral rehydration solution (ORS) with or without the inclusion of active base ingredients (carbohydrate and electrolytes). The functional ingredients included in both the control and test solutions were Melatonin in conjunction with L-theanine (Arm 1), Caffeine in conjunction with L-theanine (Arm 2), and Vitamin C in conjunction with Zinc (Arm 3), across two study periods.

The primary outcomes of this study included the relative pharmacokinetics of each functional ingredient. These included: maximum observed concentration (C max), time of maximum observed concentration (T max), cumulative Area Under the Curve (AUC) for each timepoint, (including AUC from the time of dosing to the time of last observation) and the concentration at each timepoint for the corresponding functional ingredients included in the specific study arm (i.e., melatonin, L-theanine, caffeine, vitamin C and zinc).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be healthy males or females, aged 18 to 55 inclusive at the time of screening, with a body mass index (BMI) of 18.0 to 34.9 kg/m2 (normal weight to Class I Obesity).
* Subjects must be able to understand the study, agree to the requirements and restrictions, and be willing to give voluntary consent to participate in the study.
* Subjects are willing to have up to nine (9) blood collections on a single study day. No clinically significant abnormal findings with the medical / surgical / medication history, abbreviated physical examination (vitals and Anthropometrics), or clinical laboratory investigations (blood tests) in the opinion of the Principal Investigator.
* Female subjects of childbearing potential must agree to one of the following methods of birth control from screening through the duration of the study.
* Acceptable methods include: abstinence, same-sex partner, double barrier (condom, diaphragm, or cervical cap with spermicidal foam, gel, or cream); intra-uterine device (IUD) with or without hormones in place or hormonal contraception (oral, injectable, implantable, transdermal, or vaginal) used consecutively for at least 3 month prior to screening visit; vasectomized partner or bilateral insertion of Essure® implants (or analogous) for at least 6 months prior to the screening visit; to be considered a female of non-childbearing potential, subject must have had a bilateral tubal ligation, hysterectomy or bilateral oophorectomy; or postmenopausal status with amenorrhea (no menstruation) for at least 1 year prior to the screening visit.
* Subject is willing to comply with the study restrictions.

Exclusion Criteria:

* Subjects who are participating in another Clinical Trial.
* Subjects who faint during blood collection, or who have a phobia of needles, or a phobia of blood.
* Subjects who have been diagnosed with any sleep disorder.
* Subjects who are night shift workers.
* Subjects who use tobacco or nicotine-containing products or devices within 1 year prior to the screening visit through the end of study.
* Females who are pregnant or lactating (verbal confirmation only).
* Subjects with history or presence of any clinically significant cardiovascular, pulmonary, respiratory, hepatic, renal, hematological, gastrointestinal, endocrine (e.g., insulin resistance, diabetes I or II), immunologic (e.g., arthritis), dermatologic, neurological, psychiatric disease or disorder (including anxiety or depression), or any uncontrolled medical illness which in the opinion of the Investigator would jeopardize the safety of the subject, interfere with study assessments, or impact the validity of the study results.
* Subjects with history of any gastrointestinal surgery, gastrointestinal illness which in the opinion of the Investigator would affect the digestive and absorption processes of the body (i.e., Gastric bypass, Gastroenteritis, Irritable Bowel Syndrome, Celiac Disease).
* Subjects with history of cancer (except localized skin cancer without metastases) within 5 years prior to the screening visit. Subjects who exhibit evidence of hepatic or renal dysfunction as evidenced by abnormal ALT, AST or ALP level ≥2 times of the upper limit of normal range or abnormal serum creatinine level ≥ 2.0 mg/dl or other clinically significant laboratory value per Investigator discretion.
* Subjects with positive laboratory result for HIV antibody, Hepatitis B surface antigen or Hepatitis C antibody.
* Subjects with history of substance or alcohol abuse within 1 year prior to the screening visit (whereas had to be seen in an Emergency Room, Urgent Care or was hospitalized for care of such).
* Subjects who received any investigational product within 30 days prior to the screening visit.
* Subjects with recent or current medical condition that may significantly affect the PK analysis, compromise the safety of the subject, or impact the validity of the study results in the opinion of the Investigator.
* Subjects who have a known or suspected allergy or sensitivity to study products or any of its ingredient(s) or to any comparable products in the opinion of the Investigator (e.g., caffeine, vitamin C, L-theanine (including green tea), melatonin etc.)
* Subjects who use any prescription or over-the-counter (OTC) medication, vitamins, herbal products, antacids, mineral supplements and dietary supplements, within 4 weeks prior to the 1st study period and through the end of study (with the exception of acetaminophen).
* Chronic use of NSAIDs (e.g., Ibuprofen, Advil), or use of NSAIDs at one-week prior to each study Visit.
* Subjects being treated with any known enzyme-altering drugs such as barbiturates, glucocorticoids, macrolides, antidepressants, neuroleptics, imidazole's, fluoroquinolones, calcium channel blockers, proton pump inhibitors, or H2-receptor antagonists, etc., within 30 days prior to screening or through the end of study.
* Subjects who (for whatever reason) have been on a self-restricted diet, controlled diet or special therapeutic diet, or who have had substantial changes in eating habits within 30 days prior to PK Test Period 1 or through the end of study.
* Subjects with difficulty fasting or consuming standard meals or snacks.
* Subjects with a proclivity to lose consciousness (faint / pass-out), feel weak, feel dizzy, or feel nauseous.
* Donation of blood (>300 ml) within 30 days or plasma within 7 days prior to PK Test Period 1 or through the end of study. Intolerance to venipuncture and intravenous cannulation.
* Subjects who are currently taking biotin supplements or have stopped taking Biotin within the last month to pre-study screening.
* Subjects who are currently taking or have taken within the last month before pre-study screening any form of psychoactive, or psychotropic drugs, including cannabinoids, CBD oils or THC.
* Subjects who are transgender or receiving any form of therapeutic intervention to instigate or maintain gender changes, or performance enhancing drugs, e.g., hormonal injections, steroid injections.
* Subjects who have taken L-theanine, melatonin, valerian root, GABA, tart cherry, amla, ashwagandha, rhodolia, ginseng, shatavari less than 14 days of pre-screening visit.
* Subjects whose veins have been deemed unsuitable for the study during screening checks.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Relative pharmacokinetics | 6 weeks
  The primary outcomes of this study included the relative pharmacokinetics of each functional ingredient. This included maximum observed concentration (C max) for the corresponding functional ingredients included in the specific study arm (i.e., melatonin, L-theanine, caffeine, vitamin and zinc).
Relative pharmacokinetics | 6 weeks
  The primary outcomes of this study included the relative pharmacokinetics of each functional ingredient. This included time of maximum observed concentration (T max) for the corresponding functional ingredients included in the specific study arm (i.e., melatonin, L-theanine, caffeine, vitamin C and zinc).
Relative pharmacokinetics | 6 weeks
  The primary outcomes of this study included the relative pharmacokinetics of each functional ingredient. This included: cumulative Area Under the Curve (AUC) for each timepoint, (including AUC from the time of dosing to the time of last observation) and the concentration at each timepoint for the corresponding functional ingredients included in the specific study arm (i.e., melatonin, L-theanine, caffeine, vitamin C and zinc).

CONTACTS AND LOCATIONS:
Locations (1):
- Princeton Consumer Research, Raritan, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No